CLINICAL TRIAL: NCT03417154
Title: Nivolumab and Oral Cyclophosphamide for Relapsed/Refractory Acute Myeloid Leukemia (AML) and Higher-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Nivolumab and Oral Cyclophosphamide for R/R AML and HIgh Risk MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017LS116; HM2017-33 (Other: University of Minnesota Division of Hematology, Oncology and Transplantation)
Record Dates: First submitted 2018-01-02; First posted 2018-01-31 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia; Higher Risk Myelodysplastic Syndrome
Keywords: AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Nivolumab; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Nivolumab every 2 weeks and Cyclophosphamide daily (Experimental)
  Interventions: Drug: Nivolumab; Drug: Low dose Cyclophosphamide (CTX) Daily
- Arm 2: Nivolumab every 2 weeks and Cyclophosphamide every 7 days (Experimental)
  Interventions: Drug: Nivolumab; Drug: Low dose Cyclophosphamide (CTX) Every 7 Days

INTERVENTIONS:
Drug: Nivolumab — 3mg/kg IV (or if prior alloHSCT, 1 mg/kg) over 30 minutes every 14 days on Days 1 and 15 for up to four 28-day courses.
  Other Names: Opdivo
Drug: Low dose Cyclophosphamide (CTX) Daily — Oral cyclophosphamide 50mg + nivolumab 3 mg/kg IV every 2 weeks for up to 4 courses of treatment
  Other Names: CTX
  Arms: Arm 1: Nivolumab every 2 weeks and Cyclophosphamide daily
Drug: Low dose Cyclophosphamide (CTX) Every 7 Days — Oral cyclophosphamide 350 mg every 7 days + nivolumab 3mg/kg IV every 2 weeks for up to 4 courses of treatment
  Other Names: CTX
  Arms: Arm 2: Nivolumab every 2 weeks and Cyclophosphamide every 7 days

SUMMARY:
This is a phase II trial of nivolumab and low dose cyclophosphamide (CTX) when given in combination to patients with relapsed/refractory acute myeloid leukemia (AML) and higher-risk myelodysplastic syndrome (MDS) who are not eligible for or decline hematopoietic stem cell transplant. It includes a randomized pilot sub-study during stage 1.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Meets one of the following disease criteria:

  * Primary (de novo) AML or higher-risk MDS with induction failure: No CR after 2 or more induction attempts with high dose chemotherapy or hypomethylating agents or other agents; no CR after 1 induction attempt and not eligible for a 2nd induction.. Higher risk MDS defined as risk score > 4.5 based on the revised IPSS criteria.
  * Secondary AML (from antecedent hematologic malignancy or treatment-related): Not in CR after 1 or more cycles of chemotherapy.
  * Relapsed AML: Blasts ≥5% in bone marrow or peripheral blood after prior attainment of CR; relapse at any time but currently ≥100 days following allogeneic HCT.
  * Relapsed MDS: Morphologic evidence of relapse or increase in blasts ≥5% in bone marrow or peripheral blood after prior attainment of hematologic improvement; or partial or complete response ; relapse at any time but currently ≥100 days following allogeneic HCT..
* ECOG Performance Status ≤ 2 - refer to Appendix II
* Adequate organ function within 14 days of study registration defined as:

  * Absolute Lymphocyte Count: ≥ 500 cells/mm3
  * Hepatic: total bilirubin ≤ 3 x upper limit of institutional normal (ULN); ALT and AST ≤ 5 x ULN
  * Renal: Serum creatinine ≤ 2 mg/dL
  * Pulmonary: No oxygen requirement on room air or requiring ≤ 2L supplemental O2
* Sexually active females of child bearing potential and males with partners of child bearing potential must agree to use effective contraception during therapy and continuing (23 weeks for females, 31 weeks for males) after the last dose of nivolumab
* Voluntary written consent

Exclusion Criteria:

* Pregnant or breastfeeding -The agents used in this study fall under Pregnancy Category D - Drugs which have caused, are suspected to have caused or may be expected to cause, an increased incidence of human fetal malformations or irreversible damage. Women of childbearing potential must have a negative pregnancy test (urine or serum) within 7 days of study drug administration.
* Prior allogeneic hematopoietic stem cell transplantation within previous 100 days (note patients with a prior alloHSCT receive nivolumab at the reduced dose of 1 mg/kg)
* Signs or symptoms of active graft versus host disease
* Active pneumonitis or uncontrolled infection
* Received chemotherapy drugs within previous 2 weeks
* Estimated life expectancy <28 days in the opinion of the enrolling investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona He, MD, Principal Investigator — Division of Hematology, Oncology and Transplantation, Masonic Cancer Center
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily: Nivolumab: 3mg/kg IV (or if prior alloHSCT, 1 mg/kg) over 30 minutes every 14 days on Days 1 and 15 for up to four 28-day courses.
  Low dose Cyclophosphamide (CTX): Oral cyclophosphamide 50mg + nivolumab 3 mg/kg IV every 2 weeks for up to 4 courses of treatment
- Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days: Nivolumab: 3mg/kg IV (or if prior alloHSCT, 1 mg/kg) over 30 minutes every 14 days on Days 1 and 15 for up to four 28-day courses.
  Low dose Cyclophosphamide (CTX): Oral cyclophosphamide 350 mg every 7 days + nivolumab 3mg/kg IV every 2 weeks for up to 4 courses of treatment
Period: Overall Study
Arm/Group | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Dosing Schedule of Low-dose Cyclophosphamide
Description: Number of participants with adverse events
Time Frame: 4 weeks from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days
Number analyzed (Participants) | 6 | 6
Participants | 6 | 6

2. Primary Outcome: Clinical Benefit and Immunologic Response of the Combination Therapy
Description: Overall response rate at 90 days from treatment start. Response is defined as CR + CRi + CRp + PR in AML and CR/PR/hematologic improvement (HI) in MDS.
  Complete Remission (CR) - subjects must have bone marrow regenerating normal hematopoietic cells and achieve a morphologic leukemia-free state, an ANC > 1 x 109/L and platelet count ≥ 100 x 109/L and normal marrow differential with < 5% blasts, and they will be RBC and platelet transfusion independent (defined as 1 week without RBC transfusion and 1 week without platelet transfusion). There should be no evidence of extramedullary leukemia
  Complete Remission with Incomplete Hematologic Recovery (CRi) - subjects must fulfill all the criteria for CR except for incomplete hematological recovery
  Complete Remission with Incomplete Platelet Recovery (CRp) - subjects must achieve CR except for incomplete platelet recovery
  Partial Remission (PR) - subjects must have ≥50% bone marrow blast reduction or decrease to 5 to 25%
Time Frame: 90 days from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Incidence of overall response.
Time Frame: 30 days from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Incidence of progression free survival.
Time Frame: 6 months from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Incidence of overall survival.
Time Frame: 6 months from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days
Number analyzed (Participants) | 6 | 6
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from on treatment date up until 6 months after the off treatment date, on average of 1 year.
Arm/Group | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 3/6 | 5/6
Other Adverse Events (participants affected / at risk) | 4/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily (N=6) | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days (N=6)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (3) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Nivolumab Every 2 Weeks and Cyclophosphamide Daily (N=6) | Arm 2: Nivolumab Every 2 Weeks and Cyclophosphamide Every 7 Days (N=6)
GI Disorders (Gastrointestinal disorders) | 3 (3) | 6 (15)
Edema limbs (General disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT03417154/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT03417154/ICF_001.pdf